CLINICAL TRIAL: NCT05453981
Title: A Pilot Randomized Controlled Trial on the Efficacy of Transdiagnostic Sleep and Circadian (TranS-C) Intervention on Anxiety Symptoms
Brief Title: A Pilot RCT on the Efficacy of TranS-C Intervention on Anxiety Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY024
Record Dates: First submitted 2022-07-08; First posted 2022-07-12 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Anxiety
Keywords: Anxiety; Insomnia; Transdiagnostic Sleep and Circadian Treatment; randomised controlled trial; TranS-C; Transdiagnostic Sleep intervention
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TranS-C group (Experimental): The TranS-C group will receive weekly 2 hour TranS-C group intervention delivered by 2 clinical psychology trainees for 6 weeks, contents being core modules from Harvey et al. (2016)'s protocol.
  Interventions: Behavioral: Transdiagnostic Sleep and Circadian Intervention
- CAU group (No Intervention): The CAU group will receive care as usual.

INTERVENTIONS:
Behavioral: Transdiagnostic Sleep and Circadian Intervention — Transdiagnostic Sleep and Circadian Intervention (TranS-C) integrates elements of evidence-based interventions, namely cognitive-behavioural therapy for insomnia, delayed sleep phase type, and interpersonal and social rhythm therapy. It targets common sleep disturbances in disorders and has improved disorder-focused symptoms and sleep and circadian functioning in patients with Severe mental illness (SMI).
  Arms: TranS-C group

SUMMARY:
This study will examine whether the Transdiagnostic Sleep and Circadian Intervention (TranS-C; Harvey & Buysse, 2017) can improve sleep and circadian functioning and reduce disorder-focused symptoms in patients with anxiety symptoms. Sleep disturbance is highly comorbid with GAD (Dolsen et al., 2014). TranS-C, targeting common sleep disturbances in disorders, has improved disorder-focused symptoms and sleep and circadian functioning in patients with Severe mental illness (SMI). Nonetheless, no study examined TranS-C's efficacy on GAD patients specifically. Hence, this study will be a pilot study that examines the efficacy of TranS-C on people with anxiety symptoms by comparing with a care-as-usual control group (CAU).

Around 80 Hong Kong residents aged 18 or above, with a GAD-7 score 10 or above and at least 1 sleep or circadian problem will be recruited. Eligible participants will be randomized to the TranS-C group or CAU group in a 1:1 ratio. The TranS-C group will receive 2-hour group-based TranS-C intervention delivered by clinical psychology trainees for 6 weeks under the supervision of a clinical psychologist. Both groups will complete a set of questionnaires at baseline, immediate post-treatment and 12-week follow-up. They will also complete sleep diaries throughout as homework. The outcome measures include mood, sleep, quality of life etc. This study will test whether theTranS-C intervention apparoach can be considered as a treatment for people with anxiety symptoms and sleep problems.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged ≥ 18 years;
2. Cantonese language fluency;
3. Score on GAD-7 is 10 or above (Johnson et al., 2019, Spitzer et al., 2006);
4. At least 1 sleep or circadian problem according to the Sleep and Circadian Problem Checklist, including time needed to fall asleep more than 30 minutes for more than 3 nights per week, less than 6 hours of sleep per night or at least 9 hour of sleep per night per 24 hour period for at least 3 nights per week, variability in the sleep-wake schedule at least 2.78 hours within a week, and falling asleep after 2 am on at least 3 nights per week;
5. Adequate opportunity and circumstances for sleep to occur; and willing to give informed consent and comply with the trial protocol.

Exclusion Criteria:

1. Presence of other psychiatric disorders as defined by the DSM-V diagnostic criteria;
2. Have suicidal ideation based on Beck Depression Inventory (BDI-II) Item 9 score ≥ 2;
3. Major medical or neurocognitive disorders that make participation infeasible;
4. Untreated sleep disorders based on SLEEP-50 (≥ 7 on narcolepsy; ≥ 15 on OSA; ≥ 7 on RLS/PLMD);
5. Past or current involvement in a psychological treatment programme for anxiety disorder and/or sleep problems;
6. Shift work, pregnancy, work, family, or other commitments that interfere with regular night-time sleep patterns;
7. Hospitalization;
8. A change in psychotropic drugs within 2 weeks before baseline assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Generalized Anxiety Disorder 7-item Scale (GAD-7) | baseline, immediate post-treatment and 12-week follow-up
  A brief 7-item instrument for screening for GAD and assessing its severity in clinical practice and research. Anxiety severity is categorized using scores of 5-9 (mild), 10-14 (moderate) and 15 or more (severe).

SECONDARY OUTCOMES:
Change in the Hospital Anxiety and Depression Scale (HADS) | baseline, immediate post-treatment and 12-week follow-up
  A 14-item self-rating scale that measures anxiety and depression in both hospital and community settings. It is divided into an Anxiety subscale (HADS-A) and a Depression subscale (HADS-D) both containing seven intermingled items. It is for screening purposes and not meant to be a diagnostic tool. HADS scores of 8-10, 11-14, and 15-21 represent mild, moderate, and severe anxiety and depression separately.
Change in the 7-day Consensus Sleep Diary | baseline, immediate post-treatment and 12-week follow-up
  The standardized sleep diary records sleep-onset latency (SOL; min), wake after sleep onset (WASO; min), total wake time (TWT; min), total sleep time (TST; min), time in bed (TIB; min); sleep efficiency (SE; calculated as TST/TIB * 100%), etc.
Change in the Insomnia Severity Index (ISI) | baseline, immediate post-treatment and 12-week follow-up
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
Change in the Short Form (Six-Dimension) Health Survey - The Chinese (Hong Kong) Version | baseline, immediate post-treatment and 12-week follow-up
  A preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality. The SF-6D index, scored from 0.0 (worst health state) to 1.0 (best health state).
Change in the Multidimensional Fatigue Inventory (MFI) | baseline, immediate post-treatment and 12-week follow-up
  A 20-item self-report instrument designed to measure fatigue. Ratings on a 5-point Likert scale are obtained on the dimensions of general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity. Scores on each subscale range from 4 to 20, with higher scores indicating greater fatigue.
Change in the Credibility-Expectancy Questionnaire (CEQ) | baseline, immediate post-treatment and 12-week follow-up
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success.
Change in the Insomnia Treatment Acceptability Scale (ITAS) | baseline, immediate post-treatment and 12-week follow-up
  The 8-item Insomnia Treatment Acceptability Scale (ITAS) may examine treatment acceptability. Respondents would score each item from 0 (not at all acceptable) to 4 (very acceptable) to rate if the rationale made sense, how acceptable the treatment was for them, suitability for their sleep problem, and expected effectiveness for their sleep problem.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Harvey AG, Dong L, Hein K, Yu SH, Martinez AJ, Gumport NB, Smith FL, Chapman A, Lisman M, Mirzadegan IA, Mullin AC, Fine E, Dolsen EA, Gasperetti CE, Bukosky J, Alvarado-Martinez CG, Kilbourne AM, Rabe-Hesketh S, Buysse DJ. A randomized controlled trial of the Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) to improve serious mental illness outcomes in a community setting. J Consult Clin Psychol. 2021 Jun;89(6):537-550. doi: 10.1037/ccp0000650. PMID 34264701
- [Background] Glynn LG, Valderas JM, Healy P, Burke E, Newell J, Gillespie P, Murphy AW. The prevalence of multimorbidity in primary care and its effect on health care utilization and cost. Fam Pract. 2011 Oct;28(5):516-23. doi: 10.1093/fampra/cmr013. Epub 2011 Mar 24. PMID 21436204
- [Background] Lam CL, Brazier J, McGhee SM. Valuation of the SF-6D Health States Is Feasible, Acceptable, Reliable, and Valid in a Chinese Population. Value Health. 2008 Mar-Apr;11(2):295-303. doi: 10.1111/j.1524-4733.2007.00233.x. PMID 18380642
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820